CLINICAL TRIAL: NCT05941845
Title: Study of Immunological Activity After Personalized Immunomodulatory Therapy Regulating the Th17 Pathway in Patients With Membranous Nephropathy
Brief Title: Interferon Alfa Therapy Based on Th17 Profile in Membranous Nephropathy
Acronym: ALPHAGEM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-AOIP-03
Record Dates: First submitted 2023-06-20; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Membranous Nephropathy
Keywords: Membranous nephropathy; Immunomodulatory therapy; Interferon alpha; Interleukine 17-A (IL-17A); Personalized medicine
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — peginterferon alfa-2a; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 6-month interferon alfa treatment (Experimental)
  Interventions: Drug: Peginterferon Alfa-2A 180 MCG/ML Injectable Solution

INTERVENTIONS:
Drug: Peginterferon Alfa-2A 180 MCG/ML Injectable Solution — Injections will be carried out on the Nephrology day hospitalization ward. The injections follows a personalized administration schedule: all enrolled patients will receive an injection of Pegasys® at Week 0.
  Patients with a persistent Th17 profile (cytokine profile showing IL-17A levels greater than 73 pg/ml) at Week 2 will receive a new dose of Pegasys®, followed by a monthly cytokine profile. In the case of a persistent Th17 profile, 2 injections will be given two weeks apart.
  In patients with no Th17 profile at Week 2, no Pegasys® injections will be performed at this time. Cytokine profiles will be performed monthly, and in the case of a persistent Th17 profile, 1 injection will be performed.
  In total, patients will receive a minimum of one injection and a maximum of 13 injections of 180 µg (1 injection every two weeks for 24 weeks).
  Other Names: Pegasys®, interferon alfa

SUMMARY:
Membranous Nephropathy (MN) is a renal autoimmune disease mediated by autoantibodies. Current management is based on the use of immunosuppressive therapies. MN patients with a pro-inflammatory Th17 cytokine profile have a 10.5-fold increased risk of disease relapse. Interferon-based immunomodulatory therapies are effective in blocking the production of cytokines in the Th17 pathway avoiding an increased risk of infection, unlike immunosuppressive treatments. To date, these treatments have not been evaluated in the management of MN. The aims of the ALPHAGEM project are to monitor the immunological activity of the disease before and after 6 months of personalized interferon-alfa treatment in MN patients.

DETAILED DESCRIPTION:
Membranous Nephropathy (MN) is a renal autoimmune disease mediated by autoantibodies, in particular the anti-phospholipase A2 receptor antibodies (anti-PLA2R1). The development of these autoantibodies is the consequence of a genetic predisposition, environmental factors and a dysregulation of the immune response, with increased production of pro-inflammatory Th2 and Th17 cytokines. Current management is based on the use of immunosuppressive therapies to induce immunological remission, which precedes clinical remission. Disease relapse may occur in 5-28% of patients, and may be complicated by long-term renal failure. MN patients with a pro-inflammatory Th17 cytokine profile have a 10.5-fold increased risk of disease relapse. Rituximab induces the regulatory T pathway, but has no impact on the Th17 pathway. Interferon-based immunomodulatory therapies are effective in blocking the production of cytokines in the Th17 pathway avoiding an increased risk of infection, unlike immunosuppressive treatments. These treatments have been used for many years in the management of autoimmune diseases (such as multiple sclerosis for interferon beta) and viral infectious diseases (such as chronic hepatitis B for interferon alfa), affections where the Th17 pathway plays a key pathophysiological role. To date, these treatments have not been evaluated in the management of MN. The aims of the ALPHAGEM project are to monitor the immunological activity of the disease before and after 6 months of personalized interferon-alfa treatment in MN patients with immunological relapse and a Th17-type cytokine profile, and to assess drug tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Diagnosis of membranous nephropathy PLA2R1 antibodies-mediated
3. Immunological relapse (defined as an increase in anti-PLA2R1 antibody titer > 14 RU/mL after a phase of anti-PLA2R1 antibody negativation, i.e. immunological remission)
4. Plasma IL-17A levels > 73 pg/mL after non-specific stimulation of peripheral blood immune cells
5. Symptomatic anti-proteinuric treatment at a stable, maximum-tolerated dosage;
6. Patients with: (i) a platelet count≥ 90,000 cells/mm3; (ii) a neutrophil count ≥ 1500 cells/mm3; and (iii) appropriately monitored normal thyroid function (TSH and T4) at screening

Exclusion Criteria:

1. Immunosuppressive treatment for MN in the 6 months before screening
2. Secondary MN (associated with cancer, infectious disease, autoimmune or iatrogenic disease)
3. Active nephrotic syndrome defined according to KDIGO guidelines by proteinuria > 3.5 g/day (or 3.5 g/g urine sample) and albuminemia < 30 g/L
4. Absence of previous immunological (anti-PLA2R1 antibodies < 14 RU/mL in ELISA or negative indirect immunofluorescence) and clinical (partial or complete) remission
5. Patients with a history of thrombosis or treated with anticoagulants
6. Pregnancy or breastfeeding
7. Cancer in treatment
8. Pre-existing retinopathy
9. Active and severe infections
10. Severe liver failure or cirrhosis
11. Pre-existing severe heart failure
12. Pre-existing psychiatric disorder or patient at risk of anxiety or depression (HAD Score > 11)
13. Patients who use or abuse substances
14. Hypersensitivity to active substance or excipients of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-07-24 (Estimated); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-07-24 (Estimated)

PRIMARY OUTCOMES:
Membranous nephropathy immunological activity monitoring over 6-month interferon alfa treatment | 18 months
  Intra-individual variation in anti-PLA2R1 antibody titer (ELISA titer in RU/mL), before and after 6 months of treatment with IFN alfa

SECONDARY OUTCOMES:
Nephrotic syndrome monitoring over 6-month interferon alfa treatment | Baseline to Week 24
  Intra-individual variation in proteinuria (g/g) under IFN alfa and stable symptomatic treatment
Nephrotic syndrome monitoring over 6-month interferon alfa treatment | Baseline to Week 24
  Intra-individual variation in albuminemia (g/L) under IFN alfa and stable symptomatic treatment
Immune response monitoring over 6-month interferon alfa treatment | Baseline to Week 24
  Intra-individual variation in cytokine profile (assay of 8 cytokines in pg/ml: IL-12p70; IL-17A; IL-4; IL-5; IL-1β; IL-10; IFNα; IL-6) before and after 6 months of personalized treatment with IFN alfa
Immune response monitoring over 6-month interferon alfa treatment | Baseline to Week 24
  Intra-individual variation in cytokine profile (assay of 1 cytokine in UI/ml: IFNγ) before and after 6 months of personalized treatment with IFN alfa
Clinical Tolerance monitoring over 6-month interferon alfa treatment | At Week 52
  Percentage of Participants with clinical Adverse Events (AEs)
Biological Tolerance monitoring over 6-month interferon alfa treatment | At Week 52
  Percentage of Participants with biological Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not planed